CLINICAL TRIAL: NCT01995084
Title: In Vivo Assessment of Hypoxia in Gastro-intestinal Cancer Using 18F-HX4-PET: an Optimization and Reproducibility Study
Acronym: HYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, H.W.M. van Laarhoven, M.D., Ph.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL40274.018.12
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Pancreatic Cancer; Esophageal Cancer; Rectal Cancer
Keywords: hypoxia; HX4; PET; cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Esophageal Neoplasms; Rectal Neoplasms; Hypoxia; Neoplasms | interventions — 3-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1-yl)propan-1-ol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Optimization (Experimental): Patients undergo a [F-18]HX4 PET/CT scan 2,3 and 4h after [F-18]HX4 injection.
  Interventions: Drug: [F-18]HX4
- Reproducibility (Experimental): Patients undergo two [F-18]HX4 PET/CT scans 3.5h after [F-18]HX4 injection within a 10-day time frame.
  Interventions: Drug: [F-18]HX4

INTERVENTIONS:
Drug: [F-18]HX4 — 400 MBq [F-18]HX4, is administered in a single intravenous bolus injection, followed by a saline flush.
  Other Names: [18 F]-3-Fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-; 1H-1,2,3-triazol-1-yl)propan-1-ol

SUMMARY:
Several studies have shown that tumour hypoxia may have a negative impact on the outcome of anticancer treatment. Assessment of tumor hypoxia at baseline or shortly after start of treatment may serve as a predictive marker to determine treatment efficacy at an early stage. Preferably, such an assessment is performed in vivo and non-invasively.Non-invasive imaging with positron emission tomography (PET) using the 2-nitroimidazole nucleoside analogue, 3-18F-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1- yl)propan-1-ol (18F-HX4), was tested as a new marker of tumor hypoxia. Before hypoxia-measurements can be clinically implemented for response prediction, the reproducibility of the technique should be assessed for each specific tumor type. Knowledge of reproducibility is needed to determine what change in parameters between two examinations can be considered relevant in an individual patient. Assessment of reproducibility becomes even more important in early response monitoring since the changes in the tumor induced by the treatment may be smaller during the treatment compared to response monitoring after completion of treatment. Also, as image quality of 18F-HX4-PET increases with increasing time intervals after injection, determination of the optimal time point for measurement of hypoxia is warranted.

DETAILED DESCRIPTION:
Background of the study:

Several studies have shown that tumour hypoxia may have a negative impact on the outcome of anticancer treatment. Assessment of tumor hypoxia at baseline or shortly after start of treatment may serve as a predictive marker to determine treatment efficacy at an early stage. Preferably, such an assessment is performed in vivo and non-invasively.Non-invasive imaging with positron emission tomography (PET) using the 2-nitroimidazole nucleoside analogue, 3-18F-fluoro-2-(4-((2-nitro-1H-imidazol-1-yl)methyl)-1H-1,2,3-triazol-1- yl)propan-1-ol (18F-HX4), was tested as a new marker of tumor hypoxia. Before hypoxia-measurements can be clinically implemented for response prediction, the reproducibility of the technique should be assessed for each specific tumor type. Knowledge of reproducibility is needed to determine what change in parameters between two examinations can be considered relevant in an individual patient. Assessment of reproducibility becomes even more important in early response monitoring since the changes in the tumor induced by the treatment may be smaller during the treatment compared to response monitoring after completion of treatment. Also, as image quality of 18F-HX4-PET increases with increasing time intervals after injection, determination of the optimal time point for measurement of hypoxia is warranted.

Objective of the study:

In this study, we first intend to investigate the optimal time point for measurement of hypoxia in esophageal, pancreatic and rectal cancer using 18F-HX4-PET and then assess reproducibility of hypoxia measurements in these tumor types.

Study design:

In this study two steps will be taken. 1) First, as 18F-HX4-PET image quality may improve when allowing for relatively longer time intervals after injection, in three patients with esophageal, pancreatic or rectal cancer 18F-HX4-PET scans will be performed 90, 180 and 240 minutes after injection of 18F-HX4. The time-point with the best image quality (in terms of tumor-to-background-ratio) will be chosen for the reproducibility study. 2) In the second step, patients with proven esophageal, pancreatic or rectal cancer will undergo an 18F-HX4-PET twice within one week before start of treatment. 18F-HX4-PET will be performed at 90, 180 or 240 minutes after injection of 18F-HX4, depending on the results of the first part of the study. Reproducibility of hypoxia measured by 18F-HX4-PET will be assessed. In those patients for whom tumor tissue is available which has not been treated with radiation or chemotherapy, levels of hypoxia measured by 18F-HX4-PET will be compared with endogenous hypoxia markers (HIF1-alfa, CA9, GLUT1, PAI-1, VEGF) using immunohistochemistry. In those patients that underwent 18F-HX4-PET before start of neoadjuvant treatment, levels of hypoxia measured by 18F-HX4-PET will be compared to pathological response after neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven invasive carcinoma of the esophagus, pancreas or rectum. In pancreatic cancer cytological proof or a high suspicion on CT imaging is allowed, too.
* Tumor size ≥ 1cm
* WHO-performance score 0-2
* Written informed consent

Exclusion Criteria:

* Any psychological, familial, sociological or geographical condition potentially hampering adequate informed consent or compliance with the study protocol.
* Surgery, radiation and/or chemotherapy foreseen within the timeframe needed for two PET scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Reproducibility of SUV measured with 18F-HX4 PET | Within 10 days
  Tumor SUVmean, SUVmax, Uptake Ratio
Optimal time frame between administration of 18F-HX4 and PET scan | 2-4h after injection
  Tumor SUVmean, SUVmax, Uptake Ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands